CLINICAL TRIAL: NCT06307834
Title: Restoring Grasp Ability in Stroke Survivors Through Motor Imagery-Based Training With EEG Feedback
Brief Title: Restoring Grasp Ability in Stroke Survivors Through MI-Based Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Responsible Party: Principal Investigator, Derek Kamper, Associate Professor, North Carolina State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26760; 24POST1194772 (Other Grant/Funding Number: American Heart Association (AHA))
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback - based therapy group (Experimental): In this arm/group, each participant will undergo a series of ten sessions (2-3 sessions per week) over a period of 3-5 weeks. Participants will be trained in modulating their brain activation patterns by using Mental Imagery (MI) involving various hand movements. EEG will be used to record brain responses. A visual feedback will be provided during the training to help achieve specific changes in brain responses. Once an appropriate brain response is achieved, an EMG-controlled hand exoskeleton will aid in opening and closing the hand.
  Interventions: Behavioral: Neurofeedback - based therapy
- Standard Hand exercises therapy group (Active Comparator): In this arm/group, each participant will undergo a series of ten sessions (2-3 sessions per week) over a period of 3-5 weeks. At each session, participants will practice a particular set of hand exercises. In this intervention, a variety of games, tasks, and movements will be used to improve grasping abilities. These exercises will be personalized according to each participant's interests, which will be identified through the Canadian Occupational Performance Measure and will be guided by study personnel.
  Interventions: Behavioral: Standard hand exercise therapy

INTERVENTIONS:
Behavioral: Neurofeedback - based therapy — This intervention will include mental practice of various hand movements accompanied by guided visual feedback, aimed at regulating brain activation patterns to facilitate the restoration of hand movements. We will also incorporate EMG signals to control a hand exoskeleton.
  Arms: Neurofeedback - based therapy group
Behavioral: Standard hand exercise therapy — This intervention will include engaging in a set of particular hand exercises with the aim of enhancing hand movements.
  Arms: Standard Hand exercises therapy group

SUMMARY:
Stroke is a leading cause of disability. Most stroke survivors face challenge in using their arm and hand to carry out daily task, such as grasping or holding objects. This issue makes it tough for nearly 65% of stroke survivors to return to work and take care of themselves. The cause of their disability is changes in their brain's activity patterns of the motor cortex area. Traditional therapy does not directly alter these brain changes, which makes it less effective. As a way to help stroke survivors, people are looking into ways to train the brain directly. A method they found is motor imagery, which involves mental practicing of a task. Studies suggest that this type of training can potentially alter the brain's patterns, which can be seen through EEG. An EEG shows a fixed pattern during movement, called SMR (sensory motor rhythm). Studies have found that people can learn to control this SMR through mental practice of a task. The SMR changes in a similar way during both movement and motor imagery. Therefore, mental practice of hand tasks can lead to improvement in actual hand movements. It has already been shown that stroke survivors can open their hands more easily after receiving SMR training. Along with that, they also have trouble to hold and release objects. SMR training may be able to address these issues by changing brain patterns. But it is not clear yet if SMR training can improve all three stages of grasping (open, close, release), and to what extent it can enhance overall hand function.

This study plans to include 20 adults who have experienced a stroke and have ongoing problems with moving their hands. Half of these participants will take part in a training in which they will learn to control their SMR for three distinct hand tasks (open, close, and release). The first session will be followed by eight training sessions. To guide users toward specific changes in EEG activity, we will provide visual feedback in training. As soon as an appropriate EEG change is made, a hand exoskeleton will help them open and close their hand. The other group of 10 patients will have traditional therapy. They will do 9 sessions of hand exercises. During and after the training, we will test both groups to see how well their hand function improved. The result will help us determine which training method is better for stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 - 80 years
2. Stroke-induced hand disability in one hand
3. Experienced first stroke at least 6-month prior
4. Difficulty in opening the hand & grasping objects (Stage of Hand 4 or 5 on the Chedoke-McMaster Stroke Assessment (CMSA))
5. Ability to distinguish specific shapes and colors on a computer screen

Exclusion Criteria:

1. Inability to provide informed consent
2. Suffering from severe pain in the shoulder or hand
3. Having rigid contractures in the joints of the upper limbs, or orthopedic issues that prevent joint movement
4. Presence of non-stroke neurological diseases
5. Presence of severe cognitive deficits, such as unilateral spatial neglect or aphasia
6. Experience of hand disability due to reasons other than stroke
7. Having other serious medical conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Box & Block test (BBT) | Change of value from before the intervention to immediately after the intervention
  A quick, simple and inexpensive test used to assess and monitor unilateral gross manual dexterity
Change of Action Research Arm Test (ARAT) | Change of value from before the intervention to immediately after the intervention
  A standardized measure used to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery
Change of Wolf Motor Function Test (WMFT) | Change of value from before the intervention to immediately after the intervention
  A standardized, quantitative assessment used to assess upper extremity (UE) motor ability through timed and functional tasks

CONTACTS AND LOCATIONS:
Locations (1):
- Hand Rehabilitation Lab, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the specifications and limitations outlined by the Institutional Review Boards at North Carolina State University and the University of North Carolina at Chapel Hill, behavioral and performance data will be made available to other investigators upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The deidentified data will become available after the completion of the study and remain available for three years.
Access Criteria: Data will be made available to other researchers for scientific purposes.

REFERENCES:
- [Background] Norman SL, McFarland DJ, Miner A, Cramer SC, Wolbrecht ET, Wolpaw JR, Reinkensmeyer DJ. Controlling pre-movement sensorimotor rhythm can improve finger extension after stroke. J Neural Eng. 2018 Oct;15(5):056026. doi: 10.1088/1741-2552/aad724. Epub 2018 Jul 31. PMID 30063219
- [Background] Ono T, Shindo K, Kawashima K, Ota N, Ito M, Ota T, Mukaino M, Fujiwara T, Kimura A, Liu M, Ushiba J. Brain-computer interface with somatosensory feedback improves functional recovery from severe hemiplegia due to chronic stroke. Front Neuroeng. 2014 Jul 7;7:19. doi: 10.3389/fneng.2014.00019. eCollection 2014. PMID 25071543
- [Background] Foong R, Ang KK, Quek C, Guan C, Phua KS, Kuah CWK, Deshmukh VA, Yam LHL, Rajeswaran DK, Tang N, Chew E, Chua KSG. Assessment of the Efficacy of EEG-Based MI-BCI With Visual Feedback and EEG Correlates of Mental Fatigue for Upper-Limb Stroke Rehabilitation. IEEE Trans Biomed Eng. 2020 Mar;67(3):786-795. doi: 10.1109/TBME.2019.2921198. Epub 2019 Jun 5. PMID 31180829
- [Background] Seo NJ, Rymer WZ, Kamper DG. Delays in grip initiation and termination in persons with stroke: effects of arm support and active muscle stretch exercise. J Neurophysiol. 2009 Jun;101(6):3108-15. doi: 10.1152/jn.91108.2008. Epub 2009 Apr 8. PMID 19357330